CLINICAL TRIAL: NCT07313748
Title: Palliative Care Day: Point Prevalence Survey of Palliative Care Needs in Hospitals and Residential Care Facilities for the Elderly.
Brief Title: Point Prevalence Survey of Palliative Care Needs in Hospitals and Residential Care Facilities for the Elderly.
Acronym: PCD
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 8190
Record Dates: First submitted 2025-11-21; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Palliative Care, Health Services
Keywords: PALLIATIVE CARE; unmet needs; HOSPITAL; LONG-TERM RESIDENCE

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational, point-prevalence study is to assess the burden of palliative care needs among adults hospitalised in Internal Medicine and Geriatrics wards, and among residents of long-term care facilities, on the National Palliative Care Day (11 November). The main question it aims to answer is: What is the prevalence of unmet palliative care needs in hospital and long-term care settings on 11 November? Participants (patients and residents) will be evaluated through a structured, web-based questionnaire designed for this study. The survey will collect clinical, functional, and symptom-related data- including comorbidities, mobility, nutritional status, dysphagia, pressure ulcers, indicators of palliative care needs (NECPAL), pain assessment, and delirium screening (4AT)-to produce a detailed snapshot of palliative care needs across settings.

DETAILED DESCRIPTION:
The National Palliative Care Day, held annually on 11 November, provides a unique opportunity to assess the prevalence of palliative care needs among patients in hospitals and residents of long-term care facilities. Beyond raising awareness of palliative care, this occasion supports more accurate monitoring of patients with unmet palliative needs and enables the collection of concrete data on current care provision.

This study aims to measure the prevalence of palliative care needs among adults admitted to Internal Medicine and Geriatrics wards and among residents of participating long-term care facilities on 11 November. Assessment will be performed using a purpose-designed questionnaire. The study intends to: (1) generate a detailed estimate of palliative care needs in hospital and residential settings; (2) increase awareness among healthcare professionals and promote timely identification and management of palliative care needs; and (3) highlight the relevance of a palliative approach not only in traditional palliative care services (hospice, home-based palliative care) but also within hospitals and long-term care facilities.

A point-prevalence (cross-sectional) design will be used through administration of a web-based survey.

Sample

Inclusion criteria

Participants must meet all of the following:

* age ≥18 years;
* hospitalised in participating wards or residing in participating long-term care facilities (medicalised nursing homes: RSA Medicalizzata, R2, R2D, R3) on 11 November;
* able to provide written informed consent and consent for data processing, or oral consent supported by a relative, caregiver, or proxy.

Exclusion criteria Participants will be excluded if they are unable to provide written consent or supported oral consent for participation and data processing.

Questionnaire

Palliative care needs will be assessed using a dedicated questionnaire (Appendix 1), delivered via a web platform. The instrument comprises three sections:

Facility-level data:

* region;
* ward type (Internal Medicine, Geriatrics) or care model for long-term facilities;
* number of beds and number of eligible patients;
* availability of an in-house palliative care service (hospitals) or access to specialist palliative consultation (long-term care).

Rater characteristics:

* socio-demographic data (age group, sex);
* profession, years of experience, current or completed specialty training.

Patient-level data:

* socio-demographic variables (age, sex);
* comorbidities (Charlson Comorbidity Index);
* mobility (baseline and current functional status);
* daily nutritional intake and recent decline;
* dysphagia (presence and type);
* pressure ulcers (including stage III-IV lesions);
* palliative care indicators (NECPAL);
* pain assessment (Numeric Pain Rating Scale, or PAINAD for advanced dementia);
* delirium screening (4AT).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admitted to participating Internal Medicine or Geriatrics wards or resident in participating long-term care facilities for older adults (medicalised nursing homes: RSA Medicalizzata, R2, R2D, R3) on 11 November (National Palliative Care Day)
* Able to provide: written informed consent for study participation and data processing, or oral consent supported by a relative/caregiver/legal proxy

Exclusion Criteria:

- Inability to provide written informed consent and absence of a relative/caregiver/legal proxy able to support oral consent for participation and data processing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults (≥18 years) hospitalised in Internal Medicine and Geriatrics wards, as well as residents of participating long-term care facilities for older adults (RSA Medicalizzata, R2, R2D, R3) on 11 November, the National Palliative Care Day. Participants represent a heterogeneous group of medically complex individuals, typically characterised by multimorbidity, functional impairment, advanced age, and a high burden of chronic disease. All eligible patients and residents present on the day of assessment will be considered for inclusion, provided informed consent can be obtained directly or with the support of a caregiver or legal proxy.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence | 1 DAY
  Prevalence of palliative care needs

CONTACTS AND LOCATIONS:
Overall Officials: Graziano Onder, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (2):
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma